CLINICAL TRIAL: NCT02414399
Title: Azithromycin to Prevent Post-discharge Morbidity and Mortality in Kenyan Children
Acronym: Toto Bora
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: Kenya Medical Research Institute (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Judd Walson, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00002592; R01HD079695 (NIH)
Record Dates: First submitted 2015-03-31; First posted 2015-04-10 (Estimated); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Pneumonia; Diarrhea; Malaria; Co-infection; Death; Malnutrition
Keywords: post-discharge mortality; morbidity and mortality prevention; azithromycin; linear growth
MeSH Terms: conditions — Pneumonia; Diarrhea; Malaria; Coinfection; Death; Malnutrition | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin (Experimental): Azithromycin 10mg/kg for one day, then 5mg/kg for four days, a total of five days of experimental treatment.
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): 5 days of taste/appearance/bottle-matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — oral administration of Azithromycin
  Other Names: Zithromax; Zmax
  Arms: Azithromycin
Drug: Placebo — 5 days of taste/appearance/bottle-matched inactive substance
  Arms: Placebo

SUMMARY:
Children hospitalized with severe illness in sub-Saharan Africa are at high risk of morbidity and mortality following discharge from hospital. These children represent an accessible high-risk population in which targeted interventions to prevent morbidity and mortality could have dramatic impact. A large cluster randomized trial of azithromycin delivered in a mass drug administration program within trachoma endemic areas in sub-Saharan Africa demonstrated an almost 50% mortality benefit in children 1-9 years of age in treated communities. However, mass drug administration of azithromycin leads to the rapid emergence of macrolide resistance within treated communities and is expensive. The targeted delivery of azithromycin to children at hospital discharge may be a novel and practical intervention to maximize benefit while minimizing risk of antibiotic resistance. This is a randomized, double-blind, placebo-controlled trial to determine the efficacy of azithromycin provided at discharge, compared to placebo, in reducing mortality and re-hospitalization rates in children age 1-59 months in Kenya. The study will also investigate potential mechanisms by which azithromycin may reduce morbidity and mortality in this population and will assess the emergence of antibiotic resistance among treated individuals and their primary caregivers. A cost-effectiveness analysis of the intervention will also be conducted.

DETAILED DESCRIPTION:
An estimated 3.5 million deaths occur annually in children less than 5 years of age in sub-Saharan Africa, approximately 70% of which are due to infectious causes. One-year mortality rates as high as 15% have been documented following hospital discharge in sub-Saharan Africa, a rate that is 8-fold higher than non-hospitalized children. Children being discharged from hospital in Africa may represent an accessible high-risk population in which to target interventions to reduce mortality. A recent trial of mass drug administration of azithromycin reduced childhood mortality by half among children in Ethiopia in communities receiving the intervention. However, concerns about the potential for the emergence of antimicrobial resistance, possible toxicity, and the feasibility of delivery are all barriers to community-wide distribution of antibiotics. Targeted chemotherapeutic interventions, including the use of cotrimoxazole among HIV-infected children and the use of amoxicillin or cefdinir among malnourished children, have been shown to reduce mortality in these specific vulnerable populations. Children who have been recently hospitalized are a high-risk population in which a similar targeted approach to azithromycin distribution may optimize benefit while reducing both individual and population level risks. The mechanisms by which azithromycin may impact morbidity and mortality have not been well described. Among high-risk pediatric populations with history of recent illness, azithromycin may act by treating residual disease not eliminated during inpatient therapy, by providing prophylaxis from future infectious exposures during a time of immune suppression and vulnerability following illness, by treating underlying enteric dysfunction and associated mucosal immune/gut barrier disruption and inflammation, and/or by clearing asymptomatic carriage of potentially pathogenic organisms. This is a randomized, double-blind, placebo-controlled trial of a 5-day course of azithromycin in children age 1 to 59 months discharged from hospital in Western Kenya to reduce post-discharge re-hospitalizations and mortality, to explore possible mechanisms by which azithromycin has benefit and risk, and to identify correlates and intermediate markers of re-hospitalization and death in the post discharge period.

Primary Aims Aim 1. To compare rates of re-hospitalization and mortality in the 6 months following hospital discharge among Kenyan children receiving 5-day azithromycin vs. placebo.

Hypothesis: The provision of a 5-day course of azithromycin provided at discharge will reduce hospital readmission and death within the 6 months following discharge, as compared to placebo.

Aim 2a. To evaluate possible mechanism(s) by which azithromycin may affect morbidity and mortality, by comparing reasons for re-hospitalization, prevalence of pathogen carriage, and markers of enteric dysfunction between the randomization arms.

Hypothesis: Children treated with azithromycin will experience fewer hospitalizations due to diarrhea, acute respiratory infection, and malnutrition, will be less likely to have respiratory and gastrointestinal carriage of potentially pathogenic organisms, and will have less evidence of enteric dysfunction, as compared to children treated with placebo in the 6 months following hospital discharge.

Aim 2b. To determine whether empiric administration of azithromycin at hospital discharge increases risk of antimicrobial resistance in commensal Escherichia coli (E. coli) and Streptococcus pneumoniae (S. pneumoniae) isolates from treated children and their household contacts.

Hypothesis: Isolates of commensal E. coli and S. pneumoniae from children treated with azithromycin and their household contacts will have higher levels of macrolide and β-lactam resistance, compared to the placebo group, after 90 days of follow-up, but resistance in the 2 arms will be similar by 6 months.

Aim 3. To identify correlates and intermediate markers of post-discharge mortality and hospital readmission among hospitalized Kenyan children.

Hypothesis: Children younger in age, with enteric dysfunction, higher levels of bacterial pathogen carriage,immune dysfunction, and malnutrition will experience more frequent re-hospitalizations and deaths.

Aim 4. To determine the cost-effectiveness of post-discharge administration of a 5-day course of azithromycin in settings of varying antibiotic use, re-hospitalization rates, and mortality rates.

Hypothesis: The provision of a 5-day course of azithromycin provided at discharge is cost-effective in settings with moderate to high re-hospitalization and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-59 months,
* Plan to remain in study area greater than 6 months
* Discharged from hospital following non-trauma related admission

Exclusion Criteria:

* Contraindication to azithromycin use and other prophylactic antibiotic use

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1400 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2025-12-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Judd L Walson, MD, MPH, Principal Investigator — University of Washington Department of Global Health; Patricia B Pavlinac, PhD, MS, Study Director — University of Washington Department of Global Health
Locations (1):
- Kisii Teaching and Referral Hospital, Homa Bay District Hospital, St. Paul's Mission Hospital, Kisii and Homa Bay Counties, Kenya

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for the primary analysis is available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: With publication of primary manuscript (Sep 2021)
Access Criteria: Open Access
URL: https://doi.org/10.7910/DVN/YTMFOJ

REFERENCES:
- [Background] Porco TC, Gebre T, Ayele B, House J, Keenan J, Zhou Z, Hong KC, Stoller N, Ray KJ, Emerson P, Gaynor BD, Lietman TM. Effect of mass distribution of azithromycin for trachoma control on overall mortality in Ethiopian children: a randomized trial. JAMA. 2009 Sep 2;302(9):962-8. doi: 10.1001/jama.2009.1266. PMID 19724043
- [Background] Moisi JC, Gatakaa H, Berkley JA, Maitland K, Mturi N, Newton CR, Njuguna P, Nokes J, Ojal J, Bauni E, Tsofa B, Peshu N, Marsh K, Williams TN, Scott JA. Excess child mortality after discharge from hospital in Kilifi, Kenya: a retrospective cohort analysis. Bull World Health Organ. 2011 Oct 1;89(10):725-32, 732A. doi: 10.2471/BLT.11.089235. Epub 2011 Jul 13. PMID 22084510
- [Background] Lozano R, Wang H, Foreman KJ, Rajaratnam JK, Naghavi M, Marcus JR, Dwyer-Lindgren L, Lofgren KT, Phillips D, Atkinson C, Lopez AD, Murray CJ. Progress towards Millennium Development Goals 4 and 5 on maternal and child mortality: an updated systematic analysis. Lancet. 2011 Sep 24;378(9797):1139-65. doi: 10.1016/S0140-6736(11)61337-8. Epub 2011 Sep 19. PMID 21937100
- [Background] Veirum JE, Sodeman M, Biai S, Hedegard K, Aaby P. Increased mortality in the year following discharge from a paediatric ward in Bissau, Guinea-Bissau. Acta Paediatr. 2007 Dec;96(12):1832-8. doi: 10.1111/j.1651-2227.2007.00562.x. PMID 18001338
- [Background] Snow RW, Howard SC, Mung'Ala-Odera V, English M, Molyneux CS, Waruiru C, Mwangi I, Roberts DJ, Donnelly CA, Marsh K. Paediatric survival and re-admission risks following hospitalization on the Kenyan coast. Trop Med Int Health. 2000 May;5(5):377-83. doi: 10.1046/j.1365-3156.2000.00568.x. PMID 10886803
- [Background] Keenan JD, Ayele B, Gebre T, Zerihun M, Zhou Z, House JI, Gaynor BD, Porco TC, Emerson PM, Lietman TM. Childhood mortality in a cohort treated with mass azithromycin for trachoma. Clin Infect Dis. 2011 Apr 1;52(7):883-8. doi: 10.1093/cid/cir069. PMID 21427395
- [Background] Trehan I, Goldbach HS, LaGrone LN, Meuli GJ, Wang RJ, Maleta KM, Manary MJ. Antibiotics as part of the management of severe acute malnutrition. N Engl J Med. 2013 Jan 31;368(5):425-35. doi: 10.1056/NEJMoa1202851. PMID 23363496
- [Background] Walker AS, Mulenga V, Ford D, Kabamba D, Sinyinza F, Kankasa C, Chintu C, Gibb DM; CHAP Team. The impact of daily cotrimoxazole prophylaxis and antiretroviral therapy on mortality and hospital admissions in HIV-infected Zambian children. Clin Infect Dis. 2007 May 15;44(10):1361-7. doi: 10.1086/515396. Epub 2007 Apr 12. PMID 17443476
- [Background] Roy SK, Chowdhury AK, Rahaman MM. Excess mortality among children discharged from hospital after treatment for diarrhoea in rural Bangladesh. Br Med J (Clin Res Ed). 1983 Oct 15;287(6399):1097-9. doi: 10.1136/bmj.287.6399.1097. PMID 6414583
- [Background] Wiens MO, Pawluk S, Kissoon N, Kumbakumba E, Ansermino JM, Singer J, Ndamira A, Larson C. Pediatric post-discharge mortality in resource poor countries: a systematic review. PLoS One. 2013 Jun 25;8(6):e66698. doi: 10.1371/journal.pone.0066698. Print 2013. PMID 23825556
- [Background] Berkley JA, Bejon P, Mwangi T, Gwer S, Maitland K, Williams TN, Mohammed S, Osier F, Kinyanjui S, Fegan G, Lowe BS, English M, Peshu N, Marsh K, Newton CR. HIV infection, malnutrition, and invasive bacterial infection among children with severe malaria. Clin Infect Dis. 2009 Aug 1;49(3):336-43. doi: 10.1086/600299. PMID 19548833
- [Background] Bernstein DS. Medical student indebtedness and choice of specialty. JAMA. 1992 Apr 8;267(14):1921. No abstract available. PMID 1548821
- [Background] Pavlinac PB, Singa BO, John-Stewart GC, Richardson BA, Brander RL, McGrath CJ, Tickell KD, Amondi M, Rwigi D, Babigumira JB, Kariuki S, Nduati R, Walson JL. Azithromycin to prevent post-discharge morbidity and mortality in Kenyan children: a protocol for a randomised, double-blind, placebo-controlled trial (the Toto Bora trial). BMJ Open. 2017 Dec 29;7(12):e019170. doi: 10.1136/bmjopen-2017-019170. PMID 29289941
- [Derived] Libby TE, Karani A, Tickell KD, Akech D, Singa B, Rwigi D, Kariuki K, Onamu N, Ounga D, Berkley JA, Walson JL, Scott JAG, Pavlinac PB. The effect of a 5-day course of azithromycin on Streptococcus pneumoniae carriage and antimicrobial resistance among Kenyan children discharged from hospital. J Infect Dis. 2026 Jan 16:jiag028. doi: 10.1093/infdis/jiag028. Online ahead of print. PMID 41542944
- [Derived] Atlas HE, Mogeni P, Shawon RA, Tickell KD, Bunyige L, Monchari I, Oongo S, Diakhate MM, Brander RL, Liru M, Bogonko G, Nduati R, Richardson BA, John-Stewart G, Walson JL, Singa BO, Pavlinac PB, McGrath CJ. Effect of azithromycin on post-discharge growth in Kenyan children. BMJ Glob Health. 2025 Nov 23;10(11):e020294. doi: 10.1136/bmjgh-2025-020294. PMID 41285436
- [Derived] Mogeni P, Ochieng JB, Atlas HE, Tickell KD, Rwigi D, Kariuki K, Aluoch LR, Sonye C, Apondi E, Ambila L, Diakhate MM, Singa BO, Liu J, Platts-Mills JA, Fang FC, Walson JL, Houpt ER, Pavlinac PB. Impact of Macrolide Resistance on Azithromycin for Prevention of Rehospitalization or Death Among Children Discharged From Hospitals in Western Kenya. J Infect Dis. 2025 Aug 14;232(2):e301-e308. doi: 10.1093/infdis/jiaf208. PMID 40257829
- [Derived] Pavlinac PB, Singa B, Huang ML, Shrestha L, Li V, Atlas HE, Diakhate MM, Brander R, Meshak L, Bogonko G, Tickell KD, McGrath CJ, Machuara IM, Ounga DO, Berkley JA, Richardson BA, John-Stewart G, Walson JL, Slyker J. Cytomegalovirus Viremia Predicts Postdischarge Mortality in Kenyan HIV-Exposed Uninfected Children. J Infect Dis. 2022 Nov 1;226(9):1519-1527. doi: 10.1093/infdis/jiac047. PMID 35152295
- [Derived] Pavlinac PB, Singa BO, Tickell KD, Brander RL, McGrath CJ, Amondi M, Otieno J, Akinyi E, Rwigi D, Carreon JD, Tornberg-Belanger SN, Nduati R, Babigumira JB, Meshak L, Bogonko G, Kariuki S, Richardson BA, John-Stewart GC, Walson JL. Azithromycin for the prevention of rehospitalisation and death among Kenyan children being discharged from hospital: a double-blind, placebo-controlled, randomised controlled trial. Lancet Glob Health. 2021 Nov;9(11):e1569-e1578. doi: 10.1016/S2214-109X(21)00347-8. Epub 2021 Sep 21. PMID 34559992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were withdrawn due to ineligibility (1 in the azithromycin arm and 1 in the placebo arm) therefore results are presented among 1398 instead of 1400.
Groups:
- Azithromycin (n=702): Azithromycin 10mg/kg for one day, then 5mg/kg for four days, a total of five days of experimental treatment.
  Azithromycin: oral administration of Azithromycin
- Placebo (n=696): 5 days of taste/appearance/bottle-matched placebo
  Placebo: 5 days of taste/appearance/bottle-matched inactive substance
Period: Overall Study
Arm/Group | Azithromycin (n=702) | Placebo (n=696)
Started | 702 | 696
Completed | 702 | 696
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 702 | 696 | 1398
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 18 [9 to 31] | 18 [9 to 33] | 18 [9 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276 | 294 | 570
  Male | 426 | 402 | 828
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 702 | 696 | 1398
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 702 | 696 | 1398
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 702 | 696 | 1398
Recruiting hospital [Count of Participants; unit: Participants]
  Kisii Teaching & Referral Hospital | 412 | 410 | 822
  Homa Bay County Referral Hospital | 259 | 262 | 521
  Kendu Adventist Hospital | 20 | 16 | 36
  St Paul Mission Hospital | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Re-hospitalization or Death
Description: Incidence rate of a composite outcome of mortality and hospital readmission during the 6 month post-discharge (follow-up) period.
Time Frame: 6 months
Measure: Number; unit: cases per 100 child years
Arm/Group | Azithromycin (n=702) | Placebo (n=696)
Number analyzed (Participants) | 702 | 696
cases per 100 child years
  Death or rehospitalization | 20.4 | 22.5
  Death | 4.7 | 6.0
  Rehospitalization | 18.8 | 18.6
Statistical Analysis 1: Comparison: Azithromycin (n=702) vs Placebo (n=696); Death or rehospitalization; Test type: Superiority; p = 0.58, Regression, Cox — Alpha =0.045 (to account for .005 alpha spending at interim analysis); Hazard Ratio (HR) = 0.91, 95% CI 2-sided [.64 to 1.29] — azithromycin is the numerator and placebo is the denominator
Statistical Analysis 2: Comparison: Azithromycin (n=702) vs Placebo (n=696); Death alone; Test type: Superiority; p = 0.49, Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.39 to 1.58] — Azithromycin-numerator and placebo-denominator
Statistical Analysis 3: Comparison: Azithromycin (n=702) vs Placebo (n=696); Rehospitalization alone; Test type: Superiority; p = .94, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [.70 to 1.47] — numerator-azithromycin denominator-placebo

2. Secondary Outcome: Mean Change in Length for Age Z-score (LAZ) Between Baseline and Outcome Assessment
Description: Mean change in length for age z-score (LAZ) between baseline and M3 or M6
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2024-12

3. Secondary Outcome: The Number of Children With Diarrhea Re-hospitalizations Following Randomization
Description: The number of children with diarrhea re-hospitalizations following randomization through follow-up
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2024-12

4. Secondary Outcome: The Number of Children With Acute Respiratory Illness Re-hospitalizations Following Randomization
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2024-12

5. Secondary Outcome: The Number of Children With Malnutrition Re-hospitalizations Following Randomization
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2024-12

6. Secondary Outcome: The Number of Children With Malaria Re-hospitalizations Following Randomization
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2024-12

7. Secondary Outcome: Prevalence of Enteric Pathogen Carriage
Description: Prevalence of enteric bacteria, viruses, and protozoa identified by qPCR at 3 months of follow-up
Time Frame: 3 months
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Prevalence of Streptococcus Pneumoniae Carriage
Description: Prevalence of Streptococcus pneumoniae from nasopharyngeal swabs collected at M3 and M6 follow-up timepoints.
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2024-12

9. Secondary Outcome: Number of Participants With Escherichia Coli Isolates From Fecal Samples Resistant to Azithromycin
Description: Among participants with E.coli isolated, # of participants with aizhtromycin resistance detected in E.coli form disc diffusion.
Time Frame: 6 months (E.coli isolated at baseline, month 3, and month 6)
Population: Children with E.coi isolated randomized to be in the antimicrobial resistance substudy
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 219 | 187
Participants
  M0 | 84 | 69
  M3: number analyzed (Participants) | 193 | 157
  M3 | 52 | 30
  M6: number analyzed (Participants) | 182 | 148
  M6 | 45 | 31
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; M0; Test type: Superiority — We modelled azithromycin resistance in E coli at baseline, 3 months, and 6 months of follow-up by randomisation group using generalised estimating equations with a Poisson link and exchangeable correlation structure, including site in the model. Models included an interaction term between randomisation group and follow-up timepoint (month 3 or month 6) to test whether an effect on resistance waned with time; p = 0.77, Chi-squared
Statistical Analysis 2: Comparison: Azithromycin vs Placebo; Month 3; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.088, Chi-squared
Statistical Analysis 3: Comparison: Azithromycin vs Placebo; M6; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.44, Chi-squared

10. Secondary Outcome: Proportion of Beta-lactam or Macrolide Resistance in Strep Pneumo in Children and Caregivers
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse event grade (death=grade 5, life-threatening= grade 4, severe=grade 3, moderate=grade 2, mile=grade 1) is defined according to 2014 Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events.
Arm/Group | Azithromycin (n=702) | Placebo (n=696)
All-Cause Mortality (participants affected / at risk) | 15/702 | 19/696
Serious Adverse Events (participants affected / at risk) | 52/702 | 54/696
Other Adverse Events (participants affected / at risk) | 274/702 | 276/696
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (n=702) (N=702) | Placebo (n=696) (N=696)
Grade 4 or 5 (cardiac disorders) (Cardiac disorders) | 1 | 1 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
Grade 4 or 5 congenital disorders (Congenital, familial and genetic disorders) | 0 | 1 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
Grade 4 or 5 (gastrointestinal disorders) (Gastrointestinal disorders) | 2 | 0 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
Grade 4 or 5 (general disorder) (General disorders) | 1 | 2 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
Grade 4 or 5 (infections) (Infections and infestations) | 43 | 43 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
Grade 4 or 5 (injury or poisoning) (Injury, poisoning and procedural complications) | 1 | 1 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
Grade 4 or 5 (renal & urinary disorder) (Renal and urinary disorders) | 2 | 1 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
Grade 4 or 5 (respiratory disorders) (Respiratory, thoracic and mediastinal disorders) | 3 | 3 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
Grade 4 or 5 (blood and lymphatic system disorders) (Blood and lymphatic system disorders) | 13 | 16 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
Grade 4 or 5 (nervous system disorders) (Nervous system disorders) | 1 | 5 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (n=702) (N=702) | Placebo (n=696) (N=696)
Grade 3 (not reported by system) (General disorders) | 0 | 0 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
Grade 2 (not reported by system) (General disorders) | 193 | 195 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.
Grade 1 (not reported by system) (General disorders) | 81 | 81 — Reporting all events that occurred during 6 month follow-up period. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Grades assigned using 2014 AIDS Table for Grading the Severity of Pediatric Adverse Events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT02414399/Prot_001.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT02414399/SAP_002.pdf